CLINICAL TRIAL: NCT05389254
Title: Association Between Time in Range and In-hospital Outcomes in Type 2 Diabetes Mellitus Patients With Acute Coronary Syndrome
Brief Title: Association Between Time in Range and In-hospital Outcomes in Type 2 Diabetic Patients With Acute Coronary Syndrome
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2022B034
Record Dates: First submitted 2022-05-17; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Type 2 Diabetes Mellitus; Acute Coronary Syndrome
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Acute Coronary Syndrome | interventions — Continuous Glucose Monitoring

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- real-time CGM group (Experimental): Participants in this group will be implanted with sensors of SISENSING® GS1 continuous glucose monitoring system in their left upper arm within 24 hours after hospitalization. According to the real-time CGM blood glucose data and clinical needs, researchers will carry out individualized in-hospital blood glucose standard management.
  Interventions: Device: continuous glucose monitoring system
- Capillary blood glucose monitoring group (Other): Participants in this group will be implanted with sensors of SISENSING® GS1 continuous glucose monitoring system in their left upper arm within 24 hours after hospitalization. But these patients will be blind to the CGM data. They'll receive 8-point capillary blood glucose monitoring simultaneously, which are 6am, 9am, 11am, 1pm, 4pm, 7pm, 9pm, 2am. According to the 8-point glucose data and clinical needs, researchers will carry out individualized in-hospital blood glucose standard management.
  Interventions: Device: capillary blood glucose monitoring

INTERVENTIONS:
Device: continuous glucose monitoring system — use real-time CGM system to check and adjust blood glucose
  Arms: real-time CGM group
Device: capillary blood glucose monitoring — monitor blood glucose with finger blood; real-time CGM is blind to both participants and researchers
  Arms: Capillary blood glucose monitoring group

SUMMARY:
The aim of this study is to use real-time continuous glucose monitoring (real-time CGM) system to get a 14-days blood glucose profile of the hospitalized type 2 diabetes mellitus (T2DM) patients with acute coronary syndrome (ACS), and to understand whether time in range (TIR) is associated with in-hospital outcomes of these patients. This study plans to recruit 100 patients. They will be randomly divided into 2 groups: real-time CGM group and capillary blood glucose monitoring group. All enrolled participants will receive standardized blood glucose management according to the "Expert consensus on blood glucose management of inpatients in China". The duration of the study will be 3 months. The primary endpoint is the average hospital stay and cardiac care unit (CCU) occupancy rate in T2DM patients with ACS. The secondary endpoint is a composite endpoint of nonfatal myocardial infarction, acute heart failure, heart failure rehospitalization, coronary revascularization, cardiovascular death, all-cause death.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 and ≤70 years old;
* T2DM according to 2022 American Diabetes Association standards;
* Patients admitted to hospital with either non-ST elevation acute coronary syndrome or ST-elevation myocardial infarction; coronary angiography examination data can be collected;
* a stable glucose lowering regimen for the previous 3 months;
* obtain informed consent;
* with complete clinical data.

Exclusion Criteria:

* Diagnosis of other types of diabetes, such as type 1 diabetes, gestational diabetes, secondary diabetes, etc.;
* No acute complications of diabetes, such as ketoacidosis, nonketotic hyperosmolar coma, etc.;
* Repeated severe hypoglycemia or hyperglycemia in the past 3 months;
* Patients who have had a history of allergic reactions to CGM materials or skin adhesives, alcohol or chlorhexidine disinfectants;
* Patients who have symptoms and signs of skin lesions, scarring, redness, infection or edema at the sensor application site that can affect the accuracy of sensor application or interstitial fluid glucose measurements;
* Combined with other acute disease states, such as uncontrolled severe infection, use of catecholamines or sedatives, use of ventilator, ventricular fibrillation, etc.;
* Patients who have a history of hematocrit, platelet, and hemoglobin abnormalities within past 2 months; moderate to severe anemia; or a disease (such as a coagulation disorder) that increases the risk of bleeding;
* Patients with malignant tumors, severe liver and kidney diseases, allergic diseases, mental and neurological diseases, combined with rheumatic or immune diseases;
* Using drugs that may affect blood sugar, including steroids, psychotropic drugs, anti-AIDS drugs, etc.;
* X-ray, CT, MRI examinations are scheduled during the period of wearing the sensor, and the appointment time cannot be changed to the beginning or the end of wearing;
* Patients currently participate in another clinical trial;
* Unwilling or unwilling to comply with study requirements, poor compliance, or refusal to use real time-CGM.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-06 (Estimated); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
The average hospital stay | 3 months
  The average hospital stay in hospitalized T2DM patients with ACS.
The CCU occupancy rate | 3 months
  The CCU occupancy rate in in hospitalized T2DM patients with ACS.

SECONDARY OUTCOMES:
Major adverse cardiovascular events after 3 months | 3 months
  A composite endpoint of nonfatal myocardial infarction, acute heart failure, heart failure rehospitalization, coronary revascularization, cardiovascular death, all-cause death.

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo First Hospital, Ningbo, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No